CLINICAL TRIAL: NCT01004393
Title: Phase II Trial of Subcutaneous Methylnaltrexone in the Treatment of Severe Opioid-induced Constipation in Cancer Patients
Brief Title: Methylnaltrexone for Opioid-induced Constipation in Cancer Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Vermont (Other)
Responsible Party: Principal Investigator, Steven Ades, Associate Professor, University of Vermont
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: VCC 0911; VCC 0911 (Other: Vermont Cancer Center)
Record Dates: First submitted 2009-10-28; First posted 2009-10-29 (Estimated); Results first posted 2016-02-02 (Estimated); Last update posted 2016-02-02 (Estimated); Status verified 2015-12

CONDITIONS: Neoplasms; Constipation; Opioid-Related Disorders
Keywords: Methylnaltrexone; Constipation; Narcotic Antagonists; Analgesics, Opioid; Neoplasms
MeSH Terms: conditions — Neoplasms; Constipation; Opioid-Related Disorders | interventions — methylnaltrexone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Methylnaltrexone bromide (Experimental): A single dose of methylnaltrexone will be administered subcutaneously to eligible subjects based on weight at the study entry. Since we will include subjects at all stages of cancer management, administering this study drug is considered experimental. We will use the dose approved by FDA, i.e., 0.15 mg/kg (round dose up to nearest 0.1 mL of volume) for weight less than 38 kg or greater than 114 kg; 8 mg (0.4 mL) for weight 38 kg to less than 62 kg; and 12 mg (0.6 mL) for weight 62 kg to 114 kg.
  Interventions: Drug: Methylnaltrexone bromide

INTERVENTIONS:
Drug: Methylnaltrexone bromide — Methylnaltrexone bromide, dosage based on weight (0.15 mg/kg (round dose up to nearest 0.1 mL of volume) for weight less than 38 kg or greater than 114 kg; 8 mg (0.4 mL) for weight 38 kg to less than 62 kg; and 12 mg (0.6 mL) for weight 62 kg to 114 kg), single dose
  Other Names: Relistor

SUMMARY:
The purpose of this study is to evaluate the efficacy of methylnaltrexone in relieving opioid-induced constipation in cancer patients at various stages of disease.

DETAILED DESCRIPTION:
Pain is one of the most common and important symptoms of cancer, often requiring opioid analgesics for control. However constipation is one of the most frequent and debilitating side effects of opioids, occurring in 40%-70% of patients being treated for chronic pain. Although laxatives are commonly used to manage opioid-induced constipation, these agents are not always effective or satisfactory. Methylnaltrexone bromide is a peripherally acting antagonist of the mu-opioid receptor. As a quaternary amine, the ability of methylnaltrexone to cross the blood-brain barrier is limited. This allows methylnaltrexone to function as a peripherally-acting antagonist in the gastrointestinal tract without impacting opioid-mediated analgesic effects in the central nervous system. The efficacy and safety of methylnaltrexone in treating opioid-induced constipation in patients with advanced disease receiving palliative care has been demonstrated. However the efficacy of this agent has not been evaluated in more active patients who are earlier in their disease course. The present study will evaluate the efficacy and safety of methylnaltrexone for the relief of severe opioid-induced constipation in this population and will attempt to identify factors predictive of methylnaltrexone response.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed neoplasm
* 18 years of age or older
* Have received opioids for analgesia for at least 2 weeks and been on a stable regimen of opioids and laxatives for 3 or more days before study entry
* Fewer than three laxation during the preceding week and no laxation within 24 hours before study entry, or no laxation within 48 hours before study entry
* Life expectancy of at least 6 months
* World Health Organization Performance Status 0-3
* Women of childbearing potential must have a negative pregnancy test
* Breastfeeding should be discontinued prior to study entry
* Ability to understand and the willingness to sign a written informed consent document.
* Laboratory values within a week of study entry:

Absolute neutrophil count > 1,500/microliter Hemoglobin > 7 g/dL Platelet count > 100,000/microliter Calculated calcium < 10.5 mg/dL Calculated creatinine clearance > 30 mg.min Alanine aminotransferase < 3 x upper limit of normal (ULN) Aspartate aminotransferase < 3 x ULN Alkaline phosphatase < 2.5 x ULN Bilirubin < 1.5 x ULN

Exclusion Criteria:

* Constipation not primarily caused by opioids, such as mechanical gastrointestinal obstruction or ongoing vinca alkaloid administration
* Indwelling peritoneal catheter
* Clinically active diverticular disease
* Fecal impaction
* Acute surgical abdomen
* Fecal ostomy
* Peritoneal carcinomatosis
* Known hypersensitivity to methylnaltrexone, naltrexone, or naloxone
* Administration of any investigational drug or experimental product within the previous 30 days
* Initiation of a new bowel regimen or prokinetic agents within a week of study entry

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2009-10; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Steven Ades, MD, Principal Investigator — Fletcher Allen Health Care / University of Vermont College of Medicine
Locations (1):
- Fletcher Allen Health Care, Burlington, Vermont, United States

REFERENCES:
- [Derived] Mori M, Ji Y, Kumar S, Ashikaga T, Ades S. Phase II trial of subcutaneous methylnaltrexone in the treatment of severe opioid-induced constipation (OIC) in cancer patients: an exploratory study. Int J Clin Oncol. 2017 Apr;22(2):397-404. doi: 10.1007/s10147-016-1041-6. Epub 2016 Sep 15. PMID 27628064

RESULTS

PARTICIPANT FLOW:
Groups:
- Methylnaltrexone: Methylnaltrexone bromide: Methylnaltrexone bromide, dosage based on weight (0.15 mg/kg (round dose up to nearest 0.1 mL of volume) for weight less than 38 kg or greater than 114 kg; 8 mg (0.4 mL) for weight 38 kg to less than 62 kg; and 12 mg (0.6 mL) for weight 62 kg to 114 kg), single dose
Period: Overall Study
Arm/Group | Methylnaltrexone
Started | 12
Completed | 12
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Methylnaltrexone
Number analyzed (Participants) | 12
Age, Continuous [Median (Full Range); unit: years] | 52 [27 to 87]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7
  Male | 5

OUTCOME MEASURES:

1. Primary Outcome: Rescue-free Laxation After Administration of Subcutaneous Methylnaltrexone
Time Frame: 4 hours after the dose of subcutaneous methylnaltrexone
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Methylnaltrexone
Number analyzed (Participants) | 12
percentage of participants | 33 [9.9 to 65]

2. Secondary Outcome: Laxation After Administration of Subcutaneous Methylnaltrexone
Time Frame: 24 and 48 hours after the dose of subcutaneous methylnaltrexone
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Methylnaltrexone
Number analyzed (Participants) | 12
percentage of participants
  Rescue-free Laxation within 24 hours (n=12) | 42 [15 to 72]
  Laxation within 48 hours (n=12) | 83 [52 to 98]

3. Secondary Outcome: Time to Laxation After Administration of Subcutaneous Methylnaltrexone
Time Frame: 48 hours after the dose of subcutaneous methylnaltrexone
Measure: Mean (Standard Error); unit: hours
Arm/Group | Methylnaltrexone
Number analyzed (Participants) | 12
hours
  Mean time to rescue-free laxation ≤4 hours (n=11) | 3.3 (0.134)
  Mean time to rescue-free laxation ≤24 hours (n=11) | 16 (0.155)
  Mean time to laxation ≤48 hours (n=11) | 20 (0.087)

4. Secondary Outcome: Overall Pain Scores (0-10; 0=no Pain, 10=Worst Pain) After Administration of Subcutaneous Methylnaltrexone
Time Frame: 48 hours after the dose of subcutaneous methylnaltrexone
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Methylnaltrexone
Number analyzed (Participants) | 12
units on a scale
  Average pain (0-4 hours) (n=12) | 2.9 (2.7)
  Average pain (4-24 hours) (n=12) | 2.4 (3.0)
  Average pain (24-48 hours) (n=12) | 2.3 (3.1)

5. Secondary Outcome: Symptoms of Opioid Withdrawal (Modified Himmelsbach Withdrawal Scales (Ranging 7-28 in Total; 1=None - 4=Severe for 7 Items)) After Administration of Subcutaneous Methylnaltrexone
Time Frame: 48 hours after the dose of subcutaneous methylnaltrexone
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Methylnaltrexone
Number analyzed (Participants) | 12
units on a scale
  0-4 hours (n=12) | 8.8 (1.1)
  4-24 hours (n=12) | 9.2 (2.2)
  24-48 hours (n=11) | 8.8 (1.8)

6. Secondary Outcome: Bowel Movement Assessment (Frequency, Consistency and Difficulty) After Administration of Subcutaneous Methylnaltrexone
Time Frame: 48 hours after the dose of subcutaneous methylnaltrexone
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Methylnaltrexone
Number analyzed (Participants) | 12
percentage of participants
  Frequency of ≥ 1 laxation (0-4 hours) (n=12) | 33 [9.9 to 65]
  Frequency of ≥ 1 laxation (4-24 hours) (n=12) | 42 [19 to 68]
  Frequency of ≥ 1 laxation (24-48 hours) (n=11) | 73 [43 to 90]
  Consistency (slight-very hard) (0-4 hours) (n=12) | 8 [1 to 36]
  Consistency (slight-very hard) (4-24 hours) (n=12) | 8 [1 to 36]
  Consistency (slight-very hard)(24-48 hours) (n=11) | 9 [2 to 38]
  Difficulty (severe-very severe) (0-4 hours) (n=12) | 42 [19 to 68]
  Difficulty (severe-very severe)(4-24 hours) (n=12) | 42 [19 to 68]
  Difficulty (severe-very severe)(24-48hours) (n=11) | 18 [5 to 48]

7. Secondary Outcome: Constipation Assessment (Severity and Distress) After Administration of Subcutaneous Methylnaltrexone
Time Frame: 48 hours after the dose of subcutaneous methylnaltrexone
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Methylnaltrexone
Number analyzed (Participants) | 12
percentage of participants
  Severity (severe-very severe) (0-4 hours) (n=12) | 42 [19 to 68]
  Severity (severe-very severe) (4-24 hours) (n=12) | 50 [25 to 75]
  Severity (severe-very severe) (24-48 hours) (n=11) | 27 [10 to 57]
  Distress (severe-very severe) (0-4 hours) (n=12) | 25 [9 to 54]
  Distress (severe-very severe) (4-24 hours) (n=12) | 25 [9 to 54]
  Distress (severe-very severe) (24-48 hours) (n=11) | 0 [0 to 26]

8. Secondary Outcome: Patient Satisfaction With the Study Medication After Administration of Subcutaneous Methylnaltrexone
Time Frame: 48 hours after the dose of subcutaneous methylnaltrexone
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Methylnaltrexone
Number analyzed (Participants) | 12
percentage of participants
  Satisfied-very satisfied (0-4 hours) (n=12) | 33 [14 to 61]
  Satisfied-very satisfied (4-24 hours) (n=12) | 58 [32 to 81]
  Satisfied-very satisfied (24-48 hours) (n=11) | 64 [35 to 85]
Statistical Analysis 1: Comparison: Methylnaltrexone; Test type: Superiority or Other; p = 0.161, ANOVA

ADVERSE EVENTS:
Time Frame: 4 years and 2 months
Arm/Group | Methylnaltrexone
Serious Adverse Events (participants affected / at risk) | 0/12
Other Adverse Events (participants affected / at risk) | 12/12
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Methylnaltrexone (N=12)
Abdominal pain (Gastrointestinal disorders) | 8
Flatulence (Gastrointestinal disorders) | 10
Nausea (Gastrointestinal disorders) | 9
Dizziness (Nervous system disorders) | 4
Diaphoresis (General disorders) | 7
Diarrhea (Gastrointestinal disorders) | 3
Injection site reaction (Skin and subcutaneous tissue disorders) | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No